CLINICAL TRIAL: NCT04848064
Title: A Pilot Phase I Trial of IL-21 Expanded, Off the Shelf, Third-Party Natural Killer (NK) Cells in Combination With Mogamulizumab in Patients With Cutaneous T-Cell Lymphomas or Adult T-Cell Leukemia/Lymphomas
Brief Title: Third-Party Natural Killer Cells and Mogamulizumab for the Treatment of Relapsed or Refractory Cutaneous T-cell Lymphomas or Adult T-Cell Leukemia/Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: John Reneau (Other)
Responsible Party: Sponsor-Investigator, John Reneau, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20103; NCI-2021-01375 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Adult T-Cell Leukemia/Lymphoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory Adult T-Cell Leukemia/Lymphoma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — Cyclophosphamide; fludarabine; mogamulizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (mogamulizumab, chemotherapy, NK cells) (Experimental): Patients receive mogamulizumab IV over 60 minutes on day -7 and fludarabine IV and cyclophosphamide IV on days -5 to -3. Patients receive NK cell infusion on day 0. Patients then receive mogamulizumab IV over 60 minutes on days 0, 7, 14, and 28, then every 2 weeks thereafter in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Mogamulizumab; Biological: Natural Killer Cell Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Mogamulizumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(CC Chemokine Receptor CCR4) (Human-Mouse Monoclonal KW-0761 Heavy Chain), Disulfide With Human-Mouse Monoclonal KW-0761 Kappa-Chain, Dimer; KM8761; KW-0761; Mogamulizumab-kpkc; Poteligeo
Biological: Natural Killer Cell Therapy — Given via infusion
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial is to find out the best dose, possible benefits and/or side effects of third-party natural killer cells in combination with mogamulizumab in treating patients with cutaneous T-cell lymphoma or adult T-cell leukemia/lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Immunotherapy with third-party natural killer cells, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Mogamulizumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving third-party natural killer cells in combination with mogamulizumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine safety, tolerability, and determine the maximum tolerated dose (MTD) of IL-21 expanded, off the shelf, third-party natural killer (NK) cells and mogamulizumab in patients with relapsed/refractory cutaneous T-cell lymphoma (CTCL) and adult T-cell leukemia/lymphoma (ATLL).

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR), progression free survival (PFS) and overall survival (OS) in same patient population treated with IL-21 expanded, off the shelf, third-party NK cells and mogamulizumab.

II. To determine impact of treatment on quality of life (QOL) by skindex-16 score.

CORRELATIVE OBJECTIVES:

I. To study CCR4 expression in lymphoma cells. II. To study serum cytokine levels. III. To study trafficking of third-party NK cells to skin and tissues. IV. To study the persistence of IL-21 expanded, off the shelf, third-party NK cells by chimerism studies.

OUTLINE: This is a dose-escalation study of natural killer cells.

Patients receive mogamulizumab intravenously (IV) over 60 minutes on day -7 and fludarabine IV and cyclophosphamide IV on days -5 to -3. Patients receive NK cell infusion every 2 weeks for six infusions total starting on day 0. Patients then receive mogamulizumab IV over 60 minutes on days 0, 7, 14, and 28, then every 2 weeks thereafter in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28-35 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign an informed consent form
* Age >= 18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Biopsy-proven, measurable, stage IB-IVB relapsed or refractory cutaneous T-cell lymphoma after 1 prior line of systemic therapy

  * Note: extracorporeal photopheresis will be considered a systemic therapy for this study
* Patients with large cell transformation of cutaneous T cell lymphoma are eligible
* Patients with adult T-cell leukemia/lymphoma (ATLL) of any stage and any subtypes. Patient must have had at least one standard chemotherapy and measurable disease at the time of enrollment
* Patients who relapsed after autologous or allogeneic stem cell transplant are eligible
* All cancer therapy, including radiation, topical steroid, and chemotherapy must have been discontinued at least 1 week or 3 half-lives whichever is the longest prior to treatment in this study. The only exceptions are participants who are symptomatic from their skin lesions and have been on corticosteroids for prolonged periods of time (> 60 days) without change. These patients may continue use of either systemic steroids (equivalent to < 10 mg per day of prednisone) or topical steroids if the frequency and dosage steroids has not changed for 21 days prior to the study. These participants should continue on the same dose of systemic/topical steroid throughout the study period unless they achieve a complete response at which time steroids can be tapered or discontinued. Patients are allowed to continue any medications with known activity in T cell lymphomas at the pre-enrollment doses for conditions other than T cell lymphomas (ie, steroids for sarcoidosis), as long as there is evidence of T cell lymphoma progression while patients were on these agents
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1 at study entry
* Absolute neutrophil count >= 1000/mm^3
* Platelet count >= 50,000/mm^3
* Total bilirubin =< 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and Alanine Aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x ULN

  * AST (SGOT) and ALT (SGPT) =< 5 x ULN in patients with documented hepatic involvement by lymphoma
* Calculated creatinine clearance >= 50 ml/min (by the Crockroft-Gault equation)
* Disease free of prior malignancies for >= 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast. Patients with early stage of prostate cancer under clinical surveillance without therapy are eligible. Patients with B-cell lymphomas treated with curative intent, and in remission for at least 2 years, may be in included (after discussion with principal investigator [PI])
* Negative serum pregnancy test at the time of enrollment for females of childbearing potential. Women who can get pregnant and men with partners who can become pregnant will be asked to practice a highly effective method of birth control while participating in the study that is considered medically acceptable by the study doctor.
* Life expectancy >= 90 days

Exclusion Criteria:

* Investigational therapies in the 2 weeks prior to beginning treatment on trial
* Patients with active central nervous system (CNS) involvement with lymphoma
* Patients with known human immunodeficiency virus (HIV) infection with CD4 < 350
* Patients who had solid organ transplants
* Evidence of active hepatitis B infection, based on positive surface antigen or hepatitis B deoxyribonucleic acid (DNA) polymerase chain reaction (PCR), or active hepatitis C infection based on positive PCR. Patients who are hepatitis B core antibody positive must take prophylaxis with lamivudine or equivalent and be willing to undergo monthly hepatitis B DNA PCR testing
* Present or history of progressive multifocal leukoencephalopathy (PML)
* Active grade II-IV acute or extensive chronic graft versus (vs.) host disease (GVHD)
* Patients may take steroids at any dose for disease control up to 24 hours prior to study enrollment. Steroids must have been discontinued at least 1 week or 3 half-lives whichever is the longest prior to treatment in this study, per inclusion criteria above. Topical steroids are allowed for CTCL patients
* Any illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety
* A cardiovascular disability status of New York Heart Association class >= 2
* History of severe allergic reactions to humanized monoclonal antibodies
* History of other malignancy that could affect compliance with the protocol or interpretation of results. Patients with a history of curatively treated basal or squamous cell carcinoma or Stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible. Patients with early stage of prostate cancer under clinical surveillance without therapy are eligible
* Known hypersensitivity to any of the study drugs or analogs
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior study therapy
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Recent major surgery (within 6 weeks prior to the start of study treatment) other than for diagnosis
* Receiving immunosuppressive therapy
* Prior therapy with mogamulizumab unless stopped previously for reasons other than progression or toxicity.
* Pregnant or lactating, or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to day 84
  Toxicities will be captured by Common Terminology Criteria for Adverse Events version 5. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. The incidence of severe adverse events or toxicities will be described. Will assess the proportion of patients who experience grade 3 or higher non-hematologic toxicity.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 4 months
  Will be summarized in a descriptive manner. The ORR will be calculated as the proportion of patients who achieve complete response /partial response, and provided with 95% confidence interval.
Progression free survival | From start of study treatment (from the first dose mogamulizumab [moga]) to first documentation of tumor progression (including radiographic and clinical progression) or to death due to any cause, whichever comes first, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Overall survival | From start of study treatment to date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the patient is known to be alive, whichever comes first, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Natural Killer (NK)-cell numerical expansion in vivo | Baseline to day 84
  Peripheral blood will be obtained before therapy, during the NK cell treatment period (day +42), after NK cell treatment (day +84), and at the time of progression. Donor NK-cell expansion will be defined as an absolute circulating donor-derived NK cell count that increases above the post-infusion level. Standard chimerism methods will be employed to determine origin and number of circulating NK cells.
Analysis of cytokine levels | Baseline to day 84
  Peripheral blood will be obtained before therapy, during the NK cell treatment period (day +42), after NK cell treatment (day +84), and at the time of relapse. Cytokine levels will be reported as absolute values and will be correlated with response to treatment and skindex-16 scores.
Quality of life analysis | Baseline to day 84
  Skindex-16 questionnaires will be obtained before therapy, during the NK cell treatment period (day +42), and after NK cell treatment (day +84, and every 2 months while on moga treatment). Skindex will be reported as total and specific domain scores, and described using graphical manners to show the pattern of change over treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: John C Reneau, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu